CLINICAL TRIAL: NCT01816152
Title: Phase 1 Methodology Issues in a Tailored Light Treatment for Persons With Dementia
Brief Title: Methodology Issues in a Tailored Light Treatment for Persons With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Mariana Figueiro, Professor, Population Health Science and Policy, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 20-4007; 7R01AG034157-11 (NIH)
Record Dates: First submitted 2013-03-15; First posted 2013-03-22 (Estimated); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Sleep Disturbances; Depression
Keywords: light treatment; circadian rhythms; sleep; agitation; depression
MeSH Terms: conditions — Parasomnias; Depression; Psychomotor Agitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Intervention (Active Comparator): Light levels, primary and secondary measurements are obtained after a 4-week intervention period where active lighting is experienced by patients.
  Interventions: Other: Tailored Active intervention
- Inactive intervention (Placebo Comparator): Light levels, primary and secondary measurements are obtained after a 4-week intervention period where an inactive lighting is experienced by patients
  Interventions: Other: Inactive intervention

INTERVENTIONS:
Other: Tailored Active intervention — Subjects experience a baseline for 1 week and an active intervention for 4 weeks. The active intervention is a bluish white light source delivering at least 300 lux at the eye of the patient during at least 2 hours daily.
  Arms: Active Intervention
Other: Inactive intervention — Subjects experience a baseline for 1 week and an inactive intervention for 4 weeks. The inactive intervention is a yellowish white light source delivering at most 50 lux at the eye of the patient during at least 2 hours daily.
  Arms: Inactive intervention

SUMMARY:
Tailored light treatment will increase sleep efficiency, reduce depression and reduce agitation scores in those with Alzheimer's disease and related dementia

DETAILED DESCRIPTION:
In a within subjects, randomized placebo control study, a tailored light treatment will be used for short-term (4 weeks). Outcome measures include sleep measures (actigraphy), and questionnaires probing behavior and mood in those who have been diagnosed with Alzheimer's disease and related dementia. After a 4-week washout period, a placebo control inactive light will be used for another 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate Alzheimer's disease and related dementia (ADRD)

Exclusion Criteria:

* major organ failure,
* major illness,
* history of head injury,
* hypertension or diabetes,
* use psychotropic (sleep aid) medicine, obstructing cataracts, macular degeneration, and blindness

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Sleep Disturbance | Change from Baseline (week 0) and intervention (week 4)
  Caregivers and subjects are asked to complete the Pittsburgh Sleep Quality Index (PSQI), which is assessed at baseline and after 4 weeks they are exposed to the lighting intervention. The seven component scores are summed to provide a global score ranging from 0 to 21 and a score of 5 or above indicates sleep disturbance. A higher number indications a greater sleep disturbance
Agitation | Change from Baseline (week 0) and intervention (week 4)
  Caregivers and subjects are asked to fill out the Cohen-Mansfield Agitation Score, which is assessed at baseline and after 4 weeks they are exposed to the lighting intervention. All scores are summed for one total score - a higher score indicates more agitation
Depression | Change from Baseline (week 0) and intervention (week 4)
  Caregivers and subjects are asked to fill out subjective questionnaires assessing depression using the Cornell Scale for Depression in Dementia (CSDD) Questionnaires are assessed at baseline and after 4 weeks they are exposed to the lighting intervention. The CSDD consists of 19 questions rated on a scale of 0 to 2 with all scores summed for a total score. A score greater than 12 indicates depression and a higher score indicates greater depression.

SECONDARY OUTCOMES:
Activity of Daily Living | Change from Baseline (week 0) and intervention (week 4)
  Caregivers and subjects are asked to fill out subjective Activity of Daily Living questionnaire (MDS-ADL), which is assessed at baseline and after 4 weeks they are exposed to the lighting intervention. Scores range from 4 to 18 and a higher score indicates a higher dependence.
Light/dark patterns | Change from Baseline (week 0) and intervention (week 4)
  Subjects are asked to wear a calibrated light meter to obtain light/dark and activity/rest patterns for 7 days prior to intervention and for 7 days after 3 weeks that the light treatment is applied. These data are used to determine circadian disruption (correlation between light/dark and activity/rest) and light dose.
Actigraphy | Change from Baseline (week 0) and intervention (week 4)
  Subjects are asked to wear an actigraph to obtain activity/rest patterns for 7 days prior to intervention and for 7 days after 3 weeks that the light treatment is applied. Actigraphs are used to measure sleep efficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana G Figueiro, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Icahn School of Medicine at Mount Sinai, Albany, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

REFERENCES:
- [Background] Figueiro MG, Hamner R, Higgins P, Hornick T, Rea MS. Field measurements of light exposures and circadian disruption in two populations of older adults. J Alzheimers Dis. 2012;31(4):711-5. doi: 10.3233/JAD-2012-120484. PMID 22699845
- [Background] Hanford N, Figueiro M. Light therapy and Alzheimer's disease and related dementia: past, present, and future. J Alzheimers Dis. 2013;33(4):913-22. doi: 10.3233/JAD-2012-121645. PMID 23099814
- [Result] Figueiro MG, Plitnick BA, Lok A, Jones GE, Higgins P, Hornick TR, Rea MS. Tailored lighting intervention improves measures of sleep, depression, and agitation in persons with Alzheimer's disease and related dementia living in long-term care facilities. Clin Interv Aging. 2014 Sep 12;9:1527-37. doi: 10.2147/CIA.S68557. eCollection 2014. PMID 25246779
- [Derived] Figueiro MG, Plitnick B, Roohan C, Sahin L, Kalsher M, Rea MS. Effects of a Tailored Lighting Intervention on Sleep Quality, Rest-Activity, Mood, and Behavior in Older Adults With Alzheimer Disease and Related Dementias: A Randomized Clinical Trial. J Clin Sleep Med. 2019 Dec 15;15(12):1757-1767. doi: 10.5664/jcsm.8078. Epub 2019 Nov 8. PMID 31855161